CLINICAL TRIAL: NCT03824834
Title: Morphine: a Novel Intervention to Maximize the Benefits of Exercise Training in Adults With Chronic Lung Disease and Persistent Breathlessness?
Brief Title: Morphine to Maximize the Benefits of Exercise Training in COPD or ILD and Persistent Breathlessness
Acronym: MorEx
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dennis Jensen, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Dennis Jensen, Ph.D., Associate Professor, McGill University
Organization: McGill University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MorEX_2019-5261
Record Dates: First submitted 2019-01-28; First posted 2019-01-31 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Interstitial Lung Disease
Keywords: Breathlessness; Dyspnea; Exercise; Opioids; Morphine; Exercise tolerance
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial; Dyspnea; Motor Activity | interventions — Exercise; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study medications, both morphine sulphate and placebo, will be dispensed by the research pharmacist according to the patient's randomization assignment. Neither research staff, nor patients, nor the treating physicians will be aware of the treatment assignment before or after randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise training with morphine (Experimental): Immediate-release oral morphine (syrup, 0.1 mg/kg body mass to a maximum dose of 10 mg) with supervised exercise training.
  Interventions: Drug: Exercise training with morphine
- Exercise training with placebo (Placebo Comparator): Placebo treatment with supervised exercise training.
  Interventions: Other: Exercise training with placebo

INTERVENTIONS:
Drug: Exercise training with morphine — Immediate-release oral morphine (syrup, 0.1 mg/kg body mass to a maximum dose of 10 mg) prepared in 250 mL of orange juice 30-min prior to each exercise session. Participants will complete exercise training sessions (three times per week for five weeks) on an electronically braked bike, supervised by a trained exercise specialist. Exercise sessions will be individualized based on participants' peak power output (60% PPO) determined from incremental exercise testing, and progressed to ensure the participant is exercising at a breathlessness intensity rating of between 3-5 Borg CR10 scale units and can complete at least 20-min of continuous cycling. Exercise duration will be increased in 5-min intervals up to 40-min. Thereafter, exercise intensity will be increased by 5-15% of baseline PPO.
  Arms: Exercise training with morphine
Other: Exercise training with placebo — Diluted simple syrup prepared in 250 mL of orange juice 30-min prior to each exercise session. Participants will complete exercise training sessions as per the experimental group.
  Arms: Exercise training with placebo

SUMMARY:
The purpose of this study is to explore the role of low-dose immediate-release oral morphine as a novel adjunct pharmacotherapy to enable symptomatic adults with advanced chronic obstructive pulmonary disease (COPD) or interstitial lung disease (ILD) to exercise at higher intensities for longer durations and maximize the psycho-physiological benefits of a supervised exercise training program. We hypothesize that, compared to placebo, exercise training with oral morphine will result in relatively greater improvements in exercise endurance time and intensity ratings of perceived breathlessness during constant-load cardiopulmonary cycle exercise testing (CPET) at 75% of peak power output (PPO).

DETAILED DESCRIPTION:
Supervised exercise training programs (such as pulmonary rehabilitation) are an integral component of the clinical management of COPD or ILD; a proven intervention for improving symptom burden, quality of life, emotional function, exercise capacity, and risk of hospitalization and death. While both low and high intensity exercise training benefits adults with COPD or ILD, evidence supports that higher intensity exercise training produces relatively greater physiological and symptomatic improvements. High intensity exercise of adequate duration is, however, difficult and unpleasant for people with COPD or ILD due to heightened exertional symptoms, particularly breathlessness.These symptoms persist despite the patient's underlying disease being optimally managed according to evidence-based clinical practice guideline standards.

Low-dose immediate-release oral morphine has recently shown promise as a novel adjunct therapy to reduce exertional breathlessness and increase exercise endurance time in people with advanced chronic lung disease (COPD). The purpose of this randomized, double-blind, placebo-controlled, two-arm pilot study is to further explore the role of low-dose immediate-release oral morphine as an adjunct pharmacotherapy to enable symptomatic adults with advanced COPD or ILD to exercise at higher intensities for longer durations and maximize the psycho-physiological benefits of a 5-week supervised exercise training program.

Adults with a clinical diagnosis of COPD or ILD and chronic breathlessness syndrome will be randomized in a 1:1 ratio to exercise training with oral morphine (ExT+MOR) (n=20; 10 COPD and 10 ILD) or exercise training with placebo (diluted simple syrup) (ExT+PLA) (n=20; 10 COPD and 10 ILD). All eligible participants will complete four assessment visits (Visits 1, 2, 3 and 4) and 15 exercise training (T1-15) sessions. Assessment Visits 1 and 3 will include post-bronchodilator (400 mg Salbutamol) pulmonary function testing and a symptom-limited incremental cardiopulmonary exercise test (CPET) to determine peak power output (PPO). Visits 2 and 4 will include a symptom-limited constant-load CPET at 75% of the PPO determined at Visit 1 and a dual energy x-ray absorptiometry (DEXA) scan to assess body composition. Supervised exercise training will be performed three times per week for five weeks on an electronically braked cycle ergometer, supervised by a trained exercise specialist. Exercise sessions will be individualized based on participants' pre-defined PPO (initial intensity of 60% PPO), and progressed to ensure the participant is exercising at an intensity corresponding to a breathlessness intensity rating of between 3-5 Borg 0-10 category ratio scale (CR10) units and can complete at least 20-min of continuous cycling. Exercise duration will be increased in 5-min intervals up to 40-min. Thereafter, exercise intensity will be increased by 5-15% of baseline PPO.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 35 years and over
* Clinical diagnosis of COPD or ILD
* Cigarette smoking history ≥20 years (COPD only)
* Post bronchodilator FEV1 <50% predicted and FEV1/FVC <0.70 (COPD only)
* Chronic breathlessness syndrome (modified Medical Research Council dyspnea score ≥3; Baseline Dyspnea Index focal score ≤6; and/or an Oxygen Cost Diagram rating ≤50% full scale despite optimal treatment of the underlying pathophysiology according to evidence-based clinical practice guidelines
* Report breathlessness as the main limiting factor to incremental CPET
* Body mass index >18.5 kg/m2 and <35 kg/m2

Exclusion Criteria:

* Changed respiratory medication dosage and/or frequency of administration in preceding two weeks
* Disease exacerbation/hospitalization in preceding six weeks
* Arterialized capillary CO2 tension (PacCO2) >50 mmHg at rest
* Self-reported history of drug addiction and/or substance abuse assessed with the CAIG-aid and SISAP questionnaires
* Severe excessive daytime sleepiness assessed with the Epworth Sleepiness Scale (score of 16 out of 24)
* Currently use anti-seizure and/or opioid drug(s)
* Use daytime supplemental oxygen
* Exercise-induced oxyhemoglobin desaturation to <80% on room air
* Participated in a pulmonary rehabilitation program in preceding 6 months
* Allergy/sensitivity to opioid drugs
* Significant extra-pulmonary disease that could impair exercise tolerance
* Contraindication(s) to cardiopulmonary exercise testing (e.g., significant cardiovascular, musculoskeletal, neurological disease)
* Pregnant or currently trying to become pregnant: women of child bearing potential (defined as having a menstrual period within the last 12 months) will be required to take a routine (urine) pregnancy test to rule out the possibility of pregnancy
* Self-report any of the following conditions: anemia or abnormally low blood volume; asthma; hypothyroidism; Addison's disease; renal insufficiency; hypopituitarism; severe malnutrition; digestive disease (any form of colitis disease); prostatic hypertrophy or urethral stricture
* Use of the blood thinning (anti-coagulant) drug Coumadin, Pradaxa, Xarelto and Eliquis in previous 2 weeks

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-08-06 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary exercise testing (CPET) endurance time | Immediately after exercise training program
  Cardiopulmonary exercise testing (constant-load) will be used to assess change in endurance time pre to post intervention. Endurance time will be defined as the total duration of loaded pedalling (minutes).
Borg modified 0-10 category ratio scale (Borg CR10) for breathlessness intensity | Immediately after exercise training program
  Borg modified 0-10 category ratio scale (Borg CR10) will be used to assess breathlessness intensity during constant-load CPET at isotime, defined as the highest equivalent 2-min interval of exercise completed by a given participant during each of the constant-load CPETs.

SECONDARY OUTCOMES:
Short Form Health Survey (SF-36) for quality of life | Immediately after exercise training program
  Short Form Health Survey (SF-36) will be used to assess change in quality of life pre to post intervention.
Multidimensional Dyspnoea Profile for 'usual' breathlessness | Immediately after exercise training program
  Multidimensional Dyspnoea Profile will be used to assess change in 'usual' breathlessness pre to post intervention.
Hospital Anxiety and Depression Scale (HADS) for anxiety and depressive symptoms | Immediately after exercise training program
  Hospital Anxiety and Depression Scale (HADS) will be used to assess change in anxiety and depressive symptoms pre to post intervention.
DEXA-derived body composition | Immediately after exercise training program
  DEXA will be used to assess change in fat free mass pre to post intervention. Fat free mass will be expressed as fat free mass index, which is the fat free mass per kg of total body weight per metre squared of standing height.
CPET physiological response (gas exchange) | Immediately after exercise training program
  Breath-by-breath CPET (incremental) parameters will be averaged in 30-sec intervals at rest and during exercise. The change in peak volume of oxygen consumption pre to post will be reported.
  CPET parameters will be collected over the first 30-sec period of every second minute during exercise. Three main time points will be used to evaluate exercise test parameters: (1) pre-exercise rest, defined as the steady-state period after at least 3-min of breathing on the mouthpiece while seated at rest before exercise; (2) isotime (as defined above); and (3) peak exercise, defined as the average of the last 30-sec of loaded pedaling.
CPET physiological response (power output) | Immediately after exercise training program
  Breath-by-breath CPET (incremental) parameters will be averaged in 30-sec intervals at rest and during exercise. The change in peak power output pre to post will be reported.
  CPET parameters will be collected over the first 30-sec period of every second minute during exercise. Three main time points will be used to evaluate exercise test parameters: (1) pre-exercise rest, defined as the steady-state period after at least 3-min of breathing on the mouthpiece while seated at rest before exercise; (2) isotime (as defined above); and (3) peak exercise, defined as the average of the last 30-sec of loaded pedaling.
Minimal clinically important difference breathlessness intensity | Immediately after exercise training program
  The proportion of participants meeting or exceeding the minimal clinically important difference of ≥1 Borg CR10 scale units in breathlessness intensity at isotime
Minimal clinically important difference exercise endurance | Immediately after exercise training program
  The proportion of participants meeting or exceeding the minimal clinically important difference of ≥101-sec for exercise endurance time at isotime
Safety measures - Arterialized carbon dioxide | Immediately after each treatment
  Pre to post treatment differences in arterialized carbon dioxide assessed with a blood sample from the warmed earlobe.
Safety measures - Opioid-Related Symptom Distress Scale (ORSDS) | Immediately after each treatment
  Pre to post treatment differences in ORSDS-derived measures of opioid-related side-effects
Safety measures - Adverse events | Immediately after exercise training program
  The number of participants reporting adverse events (serious and non serious).

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Jensen, Ph.D, Principal Investigator — McGill University
Locations (1):
- Montreal Chest Institute of the McGill University Health Center (MUHC), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Exercise & Respiratory Physiology Laboratory (CERPL) of McGill University — http://www.mcgill.ca/cerpl/